CLINICAL TRIAL: NCT05897853
Title: Impact of Vertigoheel® on Patients Suffering From Bilateral Vestibulopathy and Functional Dizziness in a Real-world Setting, Using PRO and QoL - a Non-interventional, Prospective, Mono-center, Observational Study
Brief Title: Impact of Vertigoheel® on Patients Suffering From Bilateral Vestibulopathy and Functional Dizziness
Acronym: HealVertigo
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Michael Strupp, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: 7564
Record Dates: First submitted 2023-05-17; First posted 2023-06-09 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Vertigo; Functional Dizziness; Bilateral Vestibulopathy
Keywords: real world evidence; non-interventional study; patient reported outcome
MeSH Terms: conditions — Vertigo; Bilateral Vestibulopathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the researcher observe how vertigo symptoms change during two months of treatment with the natural medicinal product Vertigoheel©. Adult patients suffering from vertigo symptoms can participate if they are diagnosed with bilateral vestibulopathy (BVP) or functional dizziness (FD) and assigned to Vertigoheel treatment. Participating patients receive an examination at study start and after 2 months of Vertigoheel treatment. The study focuses on patient reported outcomes assessed by questionnaires.

Vertigo symptoms are assessed by the Dizziness Handicap Inventory questionnaire. Patients' quality of life is assessed by a questionnaire. Body sway is assessed by static posturography. FD patients are additionally tested for depressive and anxiety symptoms by questionnaires. BVP patients are additionally tested for vestibular function by video head impulse test and caloric testing. Adverse events and other observations related to safety (physical examination and vital signs) are evaluated.

Vertigo is a common symptom with significant adverse effects on patients' quality of life. Regardless of the exact cause of vertigo attacks, it is important to reduce the frequency, intensity, and duration of vertigo attacks with an effective medication that has no or minimal adverse effect. Vertigoheel®, a natural medicinal product consisting of four ponderable active ingredients, is approved in Germany as treatment for vertigo of various origins. However, no systematic data are available for Vertigoheel® regarding patient-reported outcomes in BVP and FD as the most accepted endpoint in vertigo studies.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with Vertigoheel® has been chosen by the physician independently of including the patient in this non-interventional study.
* Bilateral vestibulopathy or functional dizziness according to the current diagnostic criteria of the Bárány Society
* Symptoms for > 3 months of moderate to severe intensity according to the dizziness handicap inventory [0 (minimum score) -100 (maximum score)] between 30 to 90 points.
* ≥18 years of age
* Legally competent male or female outpatient.
* Signed informed consent.
* Not pregnant (as proven by negative pregnancy test in case of woman of childbearing potential before first study drug administration) or breast-feeding.

Exclusion Criteria:

* Having taken within the last 2 months or currently taking Vertigoheel®.
* Debilitating acute or chronic illness (i.e. psychiatric illnesses).
* History of sensitivity to any component of the study drug under observation.
* Unwilling or unable to comply with all the requirements of the study protocol.
* Any relationship of dependence with the sponsor or with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients, aged ≥18 years old, diagnosed with bilateral vestibulopathy or functional dizziness were recruited from the Department of Neurology at the Hospital of the Ludwig-Maximilians-University Munich.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2022-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Strupp, Prof, MD, Principal Investigator — Department of Neurology, Ludwig-Maximilians-University Munich
Locations (1):
- Department of Neurology, Ludwig Maximilian University, Munich, Bavaria, Germany

REFERENCES:
- [Result] Ganeva D, Tiemann R, Duller S, Strupp M. Improvement of vertigo symptoms after 2 months of Vertigoheel treatment: a case series in patients with bilateral vestibulopathy and functional dizziness. Front Neurol. 2023 Oct 5;14:1264884. doi: 10.3389/fneur.2023.1264884. eCollection 2023. PMID 37869139

RESULTS

PARTICIPANT FLOW:
Groups:
- Functional Dizziness: Patients diagnosed with functional dizziness according to the current diagnostic criteria of the Bárány Society.
- Bilateral Vestibulopathy: Patients diagnosed with bilateral vestibulopathy according to the current diagnostic criteria of the Bárány Society.
Period: Overall Study
Arm/Group | Functional Dizziness | Bilateral Vestibulopathy
Started | 41 | 21
Confirmed Diagnostic Criteria at Baseline | 41 | 13
Completed | 39 | 13
Not Completed | 2 | 8
Not completed — Lost to Follow-up | 2 | 0
Not completed — Diagnostic criteria not met at baseline | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Functional Dizziness | Bilateral Vestibulopathy | Total
Number analyzed (Participants) | 41 | 13 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 5 | 24
  >=65 years | 22 | 8 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (14.9) | 64.1 (11.2) | 64.3 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 3 | 22
  Male | 22 | 10 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 41 | 13 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 41 | 13 | 54

OUTCOME MEASURES:

1. Primary Outcome: Dizziness Handicap Inventory
Description: Change from baseline in dizziness handicap inventory (DHI) after 2±1 months Vertigoheel® treatment.
  The DHI, ranging from 0 to 100 with higher scores indicating greater severity, was assessed at two time points: baseline and 2 months.
Time Frame: 2 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Functional Dizziness | Bilateral Vestibulopathy
Number analyzed (Participants) | 39 | 13
score on a scale | -12.0 [-17.8 to -6.2] | -13.2 [-19.5 to -7.0]

2. Secondary Outcome: Quality of Life (QoL)
Description: Change from baseline in quality of life (QoL) assessed by EQ-5D-5L after 2±1 months Vertigoheel® treatment.
  The EQ-5D index was used as described by Ludwig et al. (PharmacoEconomics, 2018, 36:663-74), ranging from -0.661 to 1.000, with higher scores indicating better quality of life. QoL was assessed at two time points: baseline and 2 months.
Time Frame: 2 months
Population: The QoL data were available for 31 patients with functional dizziness and 11 patients with bilateral vestibulopathy
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Functional Dizziness | Bilateral Vestibulopathy
Number analyzed (Participants) | 31 | 11
units on a scale | 0.121 [0.018 to 0.223] | 0.067 [-0.013 to 0.146]

3. Secondary Outcome: Postural Imbalance
Description: Change from baseline in body sway assessed by static posturography after 2±1 months Vertigoheel® treatment.
  Posturography was assessed as described by Brandt et al. (J Neurol 2012, 259:182-4) with an artificial neural network analysis. Category three of the method for "peripheral vestibular deficit" was evaluated for patients with bilateral vestibulopathy, and category five for "phobic postural vertigo" was evaluated for patients with functional dizziness. Posturography was assessed at two time points: baseline and 2 months. Reported values indicate the deviation from baseline values. Positive values indicate more swaying and negative values indicate less swaying. The higher the value, the more swaying (worse regulation of stand). The 2-month values were examined for significant differences from baseline values. One-sample t-Tests were used to compare mean change from baseline values versus zero (no change).
Time Frame: 2 months
Population: The postural imbalance data were available for 28 patients with functional dizziness and 13 patients with bilateral vestibulopathy
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | Functional Dizziness | Bilateral Vestibulopathy
Number analyzed (Participants) | 28 | 13
arbitrary units | 2.8 [-3.8 to 9.3] | 0.2 [-4.9 to 5.2]

4. Secondary Outcome: Depressive Symptoms in Functional Dizziness
Description: Change from baseline in depressive symptoms of functional dizziness patients assessed by PHQ-9 questionnaires after 2±1 months Vertigoheel® treatment.
  The PHQ-9, ranging from 0 to 27 with higher scores indicating greater severity, was assessed at two time points: baseline and 2 months.
Time Frame: 2 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Functional Dizziness
Number analyzed (Participants) | 39
score on a scale | -2.2 [-3.5 to -1.0]

5. Secondary Outcome: Anxiety Symptoms in Functional Dizziness
Description: Change from baseline in anxiety symptoms of functional dizziness patients assessed by GAD-7 questionnaires after 2±1 months Vertigoheel® treatment. The GAD-7, ranging from 0 to 21 with higher scores indicating greater severity, was assessed at two time points: baseline and 2 months.
Time Frame: 2 months
Population: Data from 38 patients were available for this readout.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Functional Dizziness
Number analyzed (Participants) | 38
score on a scale | -2.0 [-3.5 to -0.6]

6. Other Pre Specified Outcome: Vestibular Function in Bilateral Vestibulopathy by Video Head Impulse Test
Description: Change from baseline in vestibular function of bilateral vestibulopathy patients assessed by video head impulse test (vHIT) after 2 ± 1 months Vertigoheel ® treatment.
  The vHIT was performed as described by MacDougall et al. (Neurology, 2009, 73(14):1134-41) to evaluate the function of the vestibulo-ocular reflex (VOR) in the high frequency range for the horizontal semicircular canals.
  Based on previous HIT data from healthy, asymptomatic subjects, a normal VOR velocity gain was defined as 0.68 or greater (MacDougall et al.2009).
  Vestibular function was assessed at two time points: baseline and 2 months. Reported values indicate the deviation from baseline values. The 2-month values were examined for significant differences from baseline values. One-sample t-Tests were used to compare mean change from baseline values versus zero (no change).
Time Frame: 2 months
Population: Data from 12 patients were available for this readout.
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | Bilateral Vestibulopathy
Number analyzed (Participants) | 12
arbitrary units | -0.02 [-0.06 to 0.03]

7. Other Pre Specified Outcome: Vestibular Function in Bilateral Vestibulopathy by Caloric Testing
Description: Change from baseline in vestibular function of bilateral vestibulopathy patients assessed by caloric testing after 2 ± 1 months of Vertigoheel® treatment.
  Caloric testing was performed as described by Strupp et al. (J Vestib Res. 2017;27(4):177-89) to evaluate the function of the vestibulo-ocular reflex (VOR) in the low-frequency range of the horizontal semicircular canal on each side.
  Bilaterally reduced angular VOR function is a diagnostic criterion for bilateral vestibulopathy (BVP). Reduced caloric response, i.e., a sum of both responses per ear <6◦/sec, can be considered a safe criterion for BVP.
  Vestibular function was assessed at two time points: baseline and 2 months. Reported values indicate the deviation from baseline values. The 2-month values were examined for significant differences from baseline values. One-sample t-Tests were used to compare mean change from baseline values versus zero (no change).
Time Frame: 2 months
Population: Data from 11 patients were available for this readout.
Measure: Mean (95% Confidence Interval); unit: arbitrary units
Arm/Group | Bilateral Vestibulopathy
Number analyzed (Participants) | 11
arbitrary units | 5.5 [-4.3 to 15.3]

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Functional Dizziness | Bilateral Vestibulopathy
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/21
Other Adverse Events (participants affected / at risk) | 7/41 | 7/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Dizziness (N=41) | Bilateral Vestibulopathy (N=21)
Backache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Central retinal artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Coronavirus disease (COVID-19) (Infections and infestations) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Feeling abnormal (Nervous system disorders) | 1 (1) | 1 (1)
Injury to toe (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasia of prostate (Renal and urinary disorders) | 0 (0) | 1 (1)
Syncope (Vascular disorders) | 1 (1) | 0 (0)
Weakness of lower extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT05897853/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT05897853/SAP_001.pdf